CLINICAL TRIAL: NCT01099319
Title: Efficacy and Safety of Renalof Administration in the Treatment of Elderly Patients With Gallstones
Brief Title: Renalof in the Treatment of Elderly Patients With Gallstones
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAT-1001-CU
Record Dates: First submitted 2010-04-05; First posted 2010-04-06 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Cholelithiasis
Keywords: Dietary supplement; Renalof; gallstones; elderly
MeSH Terms: conditions — Cholelithiasis; Gallstones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renalof (Experimental)
  Interventions: Dietary Supplement: Renalof
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Renalof — One 325 mg Renalof tablet (Orally administered) every 8 hours, for 6 months.
  Arms: Renalof
Dietary Supplement: Placebo — One Placebo tablet (Orally administered) every 8 hours, for 6 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Renalof administration in the treatment of gallstones (cholelithiasis) as determined by ultrasonography and clinical evaluation in elderly patients (aged >65 years). The duration of this double-blind placebo controlled phase 3 clinical trial will be 6 months. The estimated number of patients to be recruited and randomized for the study is 40.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of cholelithiasis by ultrasonography with or without clinical symptoms.
* Signed informed consent

Exclusion Criteria:

* Previous surgical intervention for the treatment of cholelithiasis
* Cholelithiasis with acute symptoms requiring emergency surgery
* Cholelithiasis associated with neoplastic condition of any localization or origin
* Usage of other antioxidants within the duration of the clinical trial
* Handicap and/or psychiatric condition preventing treatment accomplishment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Size of calculi at month 0 and 6 (month 0 refers to the beginning of treatment and month 6 refers to the end of the treatment) | 6 month
Number of calculi at month 0 and 6 (month 0 refers to the beginning of treatment and month 6 refers to the end of the treatment) | 6 month

SECONDARY OUTCOMES:
Presence of digestive symptoms associated with cholelithiasis | 6 month
Occurrence of adverse effects during treatment | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Hernández Mojena, MD, Principal Investigator — "Dr. Salvador Allende" Clinical-Surgical-Docent Hospital
Locations (1):
- "Dr. Salvador Allende" Clinical-Surgical-Docent Hospital, Havana, La Habana, Cuba